CLINICAL TRIAL: NCT01747694
Title: The Effectiveness of Multi-respiratory Muscle Training on Respiratory Function in Patients With COPD
Brief Title: Respiratory Muscle Exercise Training in COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101-2527A3
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-10

CONDITIONS: COPD
Keywords: COPD,Respiratory muscle training,Exercise tolerance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-respiratory muscle training (Experimental): Patients will perform multi-repiratory muscle training programe for 12 weeks
  Interventions: Behavioral: Multi-respiratory muscle training
- Diaphragmatic breathing (No Intervention): Patients will be taught diaphragmatic breathing technique routinely. To practice at home lasting 12 weeks

INTERVENTIONS:
Behavioral: Multi-respiratory muscle training — Patients will be taught the diaphragmatic breathing technique at the same time also will be instructed a four-item (including upper-arm weighted exercise, body side-bends, modified sit-ups, body crunching) multi-respiratory muscle training motions. To practice three times/day, three days a week lasting 12 weeks at home.
  Arms: Multi-respiratory muscle training

SUMMARY:
COPD patients often suffer from dyspnea and exercise intolerance which lower their quality of life.The aim of this proposed study is to examine the effectiveness of multi-respiratory muscle training on respiratory function of COPD patients.

DETAILED DESCRIPTION:
The respiratory muscle training is an important part of pulmonary rehabilitation. Subjects will be recruited from the chest medicine clinic of a medical center in Northern Taiwan, randomly assigned to control and experimental groups by severity status for a 12-week muscle training intervention.The outcome measures will be performed to evaluate respiratory function, depression status and quality of life at baseline, 4, 8 and 12 weeks of training.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic Obstructive Pulmonary Disease
* Must be stable
* Never participate in respiratory muscle trainig program

Exclusion Criteria:

* Infection or acute excerbation condition
* Abdominal surgical
* Severe neuromuscular, cardiac disease or dementia

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-08 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
PE max | three months
  maximal strength of expiratory muscle

SECONDARY OUTCOMES:
PI max | three months
  maximal strength of inspiratory muscle
6MWT | three months
  six-minute walking test
MVV | three months
  maximal voluntary volume

OTHER OUTCOMES:
St. George's Respiratory Questionnaire | three months
  Disease-Specific quality of life
CES-D | three months
  assessment of depressive status

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chuan Ho, PhD, Study Chair — Chang Gung Memorial Hospital; Min-Fang Hsu, PhD student, Principal Investigator — Department of Healthcare Administration,Asia University
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan